CLINICAL TRIAL: NCT00309894
Title: Phase II Trial to Assess the Activity of Ketoconazole Plus GM-CSF in Patients With Prostate Cancer Progressive After Androgen Deprivation
Brief Title: Ketoconazole, Hydrocortisone, and GM-CSF in Treating Patients With Progressive Prostate Cancer After Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 035516; UCSF-H45860-23833-02
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sargramostim; Ketoconazole; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: sargramostim
Drug: ketoconazole
Drug: therapeutic hydrocortisone

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Drugs, such as ketoconazole, may stop the adrenal glands from making androgens. GM-CSF may help ketoconazole work better by making tumor cells more sensitive to the drug. Giving ketoconazole together with hydrocortisone and GM-CSF may be an effective treatment for prostate cancer.

PURPOSE: This phase II trial is studying how well giving ketoconazole together with hydrocortisone and GM-CSF works in treating patients with progressive prostate cancer after hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effect of ketoconazole, hydrocortisone, and sargramostim (GM-CSF) on time to clinical progression in patients with prostate cancer that has progressed on primary hormonal therapy.

Secondary

* Evaluate the objective response frequency in patients treated with this regimen.
* Investigate the safety of this regimen.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive oral ketoconazole three times daily and oral hydrocortisone twice daily on days 1-28 and sargramostim (GM-CSF) subcutaneously on days 15-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Progressive disease after androgen deprivation AND meets 1 of the following criteria:

  * Measurable disease

    * Measurable lesions ≥ 10 mm with spiral CT
    * Up to 5 lesions per organ and 10 lesions total should be identified as target lesions
  * No measurable disease

    * Patients with prostate-specific antigen (PSA)-only disease must have an elevated PSA

      * PSA evidence for progressive disease consists of a PSA level of ≥ 5 ng/mL that has risen on ≥ 2 successive occasions, ≥ 2 weeks apart
    * Patients with a positive bone scan must also have an elevated PSA
* Patients who received prior antiandrogen as a part of primary androgen ablation therapy must demonstrate disease progression after discontinuation of the antiandrogen

  * Disease progression after antiandrogen withdrawal is defined as 2 consecutive rising PSA values obtained ≥ 2 weeks apart, or documented osseous or soft tissue progression

    * Patients receiving flutamide must have had ≥ 1 of the PSA values obtained ≥ 4 weeks after flutamide discontinuation
    * Patients receiving bicalutamide or nilutamide must have had ≥ 1 of the PSA values obtained ≥ 6 weeks after antiandrogen discontinuation
* Testosterone < 50 ng/dL
* PSA ≥ 5 ng/mL

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* No serious intercurrent infections or nonmalignant uncontrolled medical illnesses
* No psychiatric illnesses OR social situations that would limit compliance
* No active or uncontrolled autoimmune disease
* ALT and AST normal
* Bilirubin normal
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit or normal (ULN)
* Hemoglobin ≥ 8 g/dL
* No other currently active malignancy except for nonmelanoma skin cancer

  * No currently active malignancy defined as therapy completed with ≤ 30% risk of relapse

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Patients must continue primary androgen deprivation therapy with a luteinizing-hormone releasing-hormone (LHRH) analogue if they have not undergone orchiectomy
* No prior systemic chemotherapy for prostate cancer

  * All other systemic chemotherapy must have been completed ≥ 2 years prior to study
* No other concurrent chemotherapy, immunotherapy, or radiotherapy
* Major surgery or radiation therapy completed ≥ 4 weeks prior to study
* No other concurrent corticosteroids, including routine use antiemetics
* No prior ketoconazole, aminoglutethimide, or corticosteroids for treatment of progressive prostate cancer
* No prior immunotherapy (e.g., vaccines or sargramostim GM-CSF)
* Patients receiving any other hormonal therapy (e.g., megestrol, finasteride, herbal product known to decrease PSA levels [e.g., saw palmetto or PC-SPES], or any systemic corticosteroid) must discontinue the agent ≥ 4 weeks prior to enrollment and progressive disease must be documented after discontinuation
* No initiation of bisphosphonate therapy within 1 month prior to starting study therapy

  * Patients on stable doses that show tumor progression are allowed to continue bisphosphonate
* No concurrent supplements or complementary medicines/botanicals, except any combination of the following:

  * Conventional multivitamin supplements
  * Selenium
  * Lycopene
  * Soy supplements
  * Vitamin E
* At least 8 weeks since prior radiopharmaceuticals (strontium chloride Sr 89, samarium Sm 153 lexidronam pentasodium)
* No other concurrent investigational or commercial anticancer agents or therapies

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-04; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to progression

SECONDARY OUTCOMES:
Response rate as measured by prostate-specific antigen and objective parameters
Frequency of grades 3-4 toxicity
Pattern of immune response as measured by immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California